CLINICAL TRIAL: NCT04276935
Title: Development of a Health-Related Symptom Index for Spanish-Speaking Persons Diagnosed With and Either Treated or Monitored for Anal High-Grade Squamous Intraepithelial Lesions (HSIL)
Brief Title: Development of a Health-Related Symptom Index for Participants With and Either Treated or Monitored for Anal High-Grade Squamous Intraepithelial Lesions
Status: Completed | Type: Observational
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Memorial Sloan Kettering Cancer Center (Other); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: AMC-A04; UM1CA121947 (NIH); U54CA137788 (NIH); NCI-2018-01740 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AMC-A04 (Other: AIDS Malignancy Consortium); AMC-A04 (Other: CTEP)
Record Dates: First submitted 2019-01-22; First posted 2020-02-19 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: High Grade Anal Canal Squamous Intraepithelial Neoplasia; Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Health Services Research (cognitive interviews): Participants take part in cognitive interviews in Spanish over 45-60 minutes.
  Interventions: Other: Interview; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Interview — Participate in cognitive interview
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial develops a health-related symptom index for participants with and either treated or monitored for anal high-grade squamous intraepithelial lesions. The health-related quality of life index may help to capture the symptoms and related experiences of living with or being treated for high-grade squamous intraepithelial lesions.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To develop a Spanish-language version of the anal cancer/high-grade squamous intraepithelial lesions outcomes research (ANCHOR) high-grade squamous intraepithelial lesions (HSIL) health-related quality of life (HRQoL) index (HQI) using state-of-the-art measure development methodology that captures the most important HRQoL symptoms and concerns of those persons diagnosed with anal HSIL and either treated or untreated for anal HSIL.

OUTLINE:

Participants take part in cognitive interviews in Spanish over 45-60 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Human immunodeficiency virus (HIV)-1 infection.
* Biopsy-proven anal HSIL within the prior nine months.
* Participant must have received anal HSIL treatment in the last nine months. If the participant's treatment plan is observation? the participant must have been diagnosed with anal HSIL in the last nine months.
* Life expectancy of greater than 5 years.
* Fluent in Spanish with limited English proficiency, per self-report.

Exclusion Criteria:

* History of anal cancer.
* Inability to understand a written consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected adult men and women with biopsy-proven anal HSIL that was treated in the last 9 months, and who are fluent in Spanish with limited English proficiency.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Atkinson, Principal Investigator — AIDS Malignancy Consortium
Locations (4):
- United States (4):
  - University of California - San Francisco, San Francisco, California
  - Jackson Memorial Hospital, Miami, Florida
  - Anal Dysplasia Clinic MidWest, Chicago, Illinois
  - Virginia Mason Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Spanish-speaking ANCHOR Participants: Participants were eligible if they were Spanish-speaking with limited English proficiency and had been diagnosed with anal high-grade squamous intraepithelial lesions in the prior nine months.
Period: Overall Study
Arm/Group | Spanish-speaking ANCHOR Participants
Started | 20
Round 1 | 10
Round 2 | 7
Completed | 17
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: Spanish Speaking ANCHOR Participants
Groups:
- Spanish-speaking ANCHOR Participants: Participants were eligible if they were ...
Arm/Group | Spanish-speaking ANCHOR Participants
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 52 [36 to 68]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender Identification: Cisgender Male | 12
  Gender Identification: Cisgender Female | 3
  Gender Identification: Transgender Female | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Development of Spanish-language Version of the Anal Cancer/High-grade Squamous Intraepithelial Lesions (HSIL) Outcomes Research (ANCHOR) Health-related Quality of Life (HRQoL) Index-Round 1 and Round 2
Description: Participants completed A-HRSI, as aurally administered over telephone to indicate whether there were any items or aspects of the instructions that were difficult to understand, and then complete a process of retrospective probing. Summary reports from the Round 1 interview were coded to highlight any instances where a participant indicated that they experienced difficulty with an item or concept within an item. For any item that was reported by at least three participants as difficult for any reason, that item or concept was reviewed to determine whether the difficulty was due to (1) the concept being measured or (2) a translation issue (i.e., register, jargon, or regionalism). These items were revised during a research team panel discussion and used in Round 2 interviews with additional eligible participants. A similar process was used for Round 2.
Time Frame: 45-60 minutes during the telephone call in each round.
Population: Round 1 included 10 participants and Round 2 had 7 respondents. The Number Analyzed in the Rows differs based on the round of the interview during which the response was recorded.
Measure: Number; unit: participants
Groups:
- Spanish Speaking ANCHOR Participants: Participants take part in cognitive interviews in Spanish over 45-60 minutes.
  Interview: Participate in cognitive interview
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
Arm/Group | Spanish Speaking ANCHOR Participants
Number analyzed (Participants) | 17
participants
  R1 Difficulty with "quite a bit (bastante" and "very much" (mucho)": number analyzed (Participants) | 10
  R1 Difficulty with "quite a bit (bastante" and "very much" (mucho)" | 4
  R2 difficulty with "not at all (para nada)" and "not applicable": number analyzed (Participants) | 7
  R2 difficulty with "not at all (para nada)" and "not applicable" | 3
  R1 difficulty understanding the noun "defecación" (defecate/defecating): number analyzed (Participants) | 10
  R1 difficulty understanding the noun "defecación" (defecate/defecating) | 3
  R1 "debres personales" is unclear and does not relate to the daily care activities used as example: number analyzed (Participants) | 10
  R1 "debres personales" is unclear and does not relate to the daily care activities used as example | 3
  R2 "Movilzarse" is not specific enough to the act of physical movement (e.g., walking): number analyzed (Participants) | 7
  R2 "Movilzarse" is not specific enough to the act of physical movement (e.g., walking) | 3
  R2 Term "tareas" is confusing: number analyzed (Participants) | 10
  R2 Term "tareas" is confusing | 3
  R2 the example "hacer la colada" was characterized as "too regional" or "unfamiliar": number analyzed (Participants) | 10
  R2 the example "hacer la colada" was characterized as "too regional" or "unfamiliar" | 3
  R2 term "ocio" was viewed by three participants as an "archaic" phrase for "leisure": number analyzed (Participants) | 10
  R2 term "ocio" was viewed by three participants as an "archaic" phrase for "leisure" | 3

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed.
Arm/Group | Spanish-speaking ANCHOR Participants
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2022-11-08): https://cdn.clinicaltrials.gov/large-docs/35/NCT04276935/Prot_000.pdf